CLINICAL TRIAL: NCT03256981
Title: Targeted Therapy With or Without Dose Intensified Radiotherapy for Oligo-progressive Disease in Oncogene-addicted Lung Tumours
Brief Title: Stereotactic Body Radiotherapy for the Treatment of OPD
Acronym: HALT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2016/10061
Record Dates: First submitted 2017-08-10; First posted 2017-08-22 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: NSCLC
Keywords: SBRT; Oligoprogressive disease; NSCLC; TKI
MeSH Terms: interventions — Radiosurgery; Tyrosine Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT and continued TKI therapy (Experimental): Patients will continue to receive background TKI treatment as prior to trial entry.
  Simultaneous administration (SBRT & TKI) or break in TKI during SBRT will be by centre preference and determined prior to commencing recruitment.
  Repeat SBRT will be permissible upon development of subsequent OPD lesions dependent on SBRT suitability and total progression lesion number at any one point remaining ≤ 5.
  Interventions: Radiation: SBRT
- Continued TKI therapy alone (Active Comparator): Continuation on the same background TKI treatment as prior to trial entry
  Interventions: Drug: TKI

INTERVENTIONS:
Radiation: SBRT — SBRT dose and fractionation dependent on site of metastasis and proximity to critical normal tissues.
  Other Names: Stereotactic body radiotherapy; SABR
  Arms: SBRT and continued TKI therapy
Drug: TKI — Continued background TKI alone
  Other Names: Tyrosine Kinase Inhibitor
  Arms: Continued TKI therapy alone

SUMMARY:
HALT is a phase II, randomised multi-centre study with integrated seamless continuation to phase III trial following acceptable safety and feasibility assessment.

HALT aims to recruit 110 patients with mutation positive advanced NSCLC with oligoprogressive disease (OPD) following initial response to a Tyrosine Kinase Inhibitor (TKI).

DETAILED DESCRIPTION:
Eligible patients will be randomised to receive either SBRT or no SBRT at a ratio of 2:1 (SBRT : no SBRT), with all patients continuing to receive background treatment with TKI therapy as clinically indicated and as per standard care. Patients randomised to receive SBRT will receive a dose and fractionation schedule dependent on OPD lesion site and proximity to critical normal tissues. All patients will be seen 8 weeks post randomisation, then 3 monthly in line with routine care.

HALT aims to assess whether in patients with mutation positive advanced NSCLC the use of SBRT to ≤ 3 sites of OPD with continuation of TKI improves progression-free survival (PFS) compared with continuation of TKI alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 16 years of age
2. Established histological diagnosis of advanced NSCLC, not suitable for radical treatment, with defined actionable mutation receiving targeted TKI therapy
3. Clinical and/or radiologically confirmed response to TKI therapy (assessed locally usually 2-3 months post commencing TKI)
4. Confirmed OPD defined as ≤ 5 extracranial sites of progressive disease. All sites must be visible, imaging defined targets and suitable for treatment with SBRT as determined by the virtual multi-disciplinary team (MDT) and in accordance with the HALT Radiotherapy planning and delivery guidance document.
5. Adequate baseline organ function to allow SBRT to all relevant targets
6. Predicted life expectancy ≥ 6 months
7. Karnofsky Index ≥ 60% and ECOG 0-2
8. Provision of written informed consent

Exclusion Criteria:

1. > 5 extracranial sites of progressive disease
2. Progressing or newly diagnosed brain metastases identified at the time of trial entry, not amenable to radical surgery or SRS. Previously treated brain metastases (i.e palliative radiotherapy or systemic therapy) which have remained clinically and radiologically stable for ≥ 6 months are permissible.
3. Prior radiotherapy near the oligoprogressive lesion precluding ablative SBRT. Suitability of lesions for ablative SBRT as part of the trial defined in section 4.1 of this document and will be determined by the HALT virtual MDT
4. Co-morbidities considered clinically precluding the safe use of SBRT (as detailed in the HALT radiotherapy planning and delivery guidelines).
5. Any psychological, sociological or geographical issue potentially hampering compliance with the study
6. Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Time from randomisation to the first of one of the above events or death. Assessed 8 weeks post-randomisation and 3-monthly thereafter (up to 24 months)
  The primary outcome measure is progression free survival defined as the time from randomisation to the first of one of the following events or death from any cause:
  * Clinically symptomatic progression requiring palliative tumour-specific oncological intervention (e.g. change in systemic therapy or localised non-SBRT radiotherapy) as determined by the treating physician.
  * New or existing intra-cranial lesions not amenable to radical surgery or Stereotactic radiosurgery (SRS).
  * Development of new extra-cranial lesions or progression of existing extra-cranial lesions not meeting the criteria for
  * SBRT treatment (e.g. size >7cm)
  * Development of >5 new or progressing extra-cranial lesion at any one point in time (i.e. widespread progression)

SECONDARY OUTCOMES:
Time to next line of systemic therapy or palliative care | Time from randomisation to change in therapy or referral to palliative care due to clinical progression as determined by the treating physician, or death. Assessed 3-monthly until progression and 6-monthly thereafter (up to 24 months).
Overall survival | Time from randomisation until death from any cause. Assessed up to 24 months.
Patterns of disease progression identified from CT scans to further document natural history of oncogene-addicted NSCLC | Assessed 3-monthly up to 24 months.
Radiotherapy toxicities (acute events) | Baseline, 8 weeks and 3-monthly intervals during follow-up (a minimum of 6 months).
  Acute events are defined as ≤ 90 days post SBRT start date (applicable for each subsequent course of SBRT where relevant) assessed using CTCAE v4.0.
Radiotherapy toxicities (late events) | Baseline, 8 weeks and 3-monthly intervals during follow-up (a minimum of 6 months).
  Late events are defined as > 90 days post SBRT start date (applicable for each subsequent course of SBRT where relevant) assessed using CTCAE v4.0.
Quality of Life (EQ-5D-5L) | Baseline, 8 weeks and at the first 3 month visit.
  Assessed using EQ-5D-5L
Quality of Life (EORTC QLQ-C30) | Baseline, 8 weeks and at the first 3 month visit.
  Assessed using EORTC QLQ-C30
Measurement of resistant sub-clones in Circulating tumour DNA (ctDNA) | Baseline, 8 weeks post-randomisation and 3-monthly intervals during follow-up (up to 24 months).
Time to failure of next line treatment | Time from randomisation to disease progression on next line of active systemic therapy. Assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona McDonald, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (29):
- France (2):
  - Institut Gustave Roussy, Paris
  - Institut Claudius Régaud, Toulouse
- Italy (2):
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Ospedale San Luigi Gonzaga - Universita Di Torino, Torino
- Spain (3):
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - University Hospital Virgen del Rocio, Seville
- Switzerland (4):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Hopital Cantonal Universitaire De Geneve, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitatsSpital Zurich, Zurich
- United Kingdom (18):
  - Royal Marsden Hosital, Sutton, England
  - Royal Marsden Hospital, Chelsea, London
  - Royal Surrey County Hospital, Guildford, Surrey
  - Belfast City Hospital, Belfast
  - Bristol Haematology and Oncology Centre, Bristol
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Castle Hill Hospital, Hull
  - Leicester Royal Infirmary, Leicester
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Guy's Hospital, London
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Lee J, Koom WS, Byun HK, Yang G, Kim MS, Park EJ, Ahn JB, Beom SH, Kim HS, Shin SJ, Kim K, Chang JS. Metastasis-Directed Radiotherapy for Oligoprogressive or Oligopersistent Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2022 Jun;21(2):e78-e86. doi: 10.1016/j.clcc.2021.10.009. Epub 2021 Nov 18. PMID 34903471